CLINICAL TRIAL: NCT02786030
Title: Integrated Primary Care for Chronic Lung Diseases in Less Developed Countries: Pragmatic Trial of the Practical Approach to Care Kit in Brazil (PACK Brazil)
Brief Title: Integrated Primary Care for Chronic Lung Disease: PACK Brazil
Acronym: PACKBrazilR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other); Santa Catarina Federal University (Other); University of Cape Town (Other); Federal University of Bahia (Other); Medical Research Council, South Africa (Other); University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PACKBrazil1
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Doctors and nurses in each clinic will receive printed copies of the patient management tool (PMT) and outreach education training. First trainers will be trained, then trainers will train groups of doctors and nurses at their workplaces, showing them how to use the guidelines, and using their own patients and clinical problems as examples. This outreach training is repeated several times in short sessions.
  Interventions: Behavioral: Outreach education training
- Control (Active Comparator): Doctors and nurses in each clinic will receive printed copies of the patient management tool (PMT) but will not receive outreach education training.
  Interventions: Behavioral: No outreach education training

INTERVENTIONS:
Behavioral: Outreach education training — Printed copies of the patient management tool (PMT) and outreach education training
  Arms: Intervention
Behavioral: No outreach education training — Printed copies of the patient management tool (PMT) without outreach education training
  Arms: Control

SUMMARY:
This study will evaluate a complex intervention based on a patient management tool (PMT), combined with educational outreach to primary care doctors, nurses and other health workers, in the Brazilian city of Florianopolis. The intervention is aimed at improving the quality of respiratory care and respiratory health outcomes, and comorbid conditions, in adults with asthma and chronic obstructive pulmonary disease (COPD). The effectiveness of the intervention will be assessed by randomly allocating 48 primary care clinics to receive the intervention or not, and comparing patient and clinic level endpoints that reflect the health and quality of care provided over the following year. About 1250 patients known to have been diagnosed with asthma and 700 with COPD in participating clinics and will be included in the study. The primary endpoints for patients with asthma and COPD, respectively, will be composite scores indicating appropriate prescribing and diagnostic testing. The third primary endpoint, among all adult clinic users, will be rates of new diagnoses of asthma and COPD in each clinic. Secondary endpoints will include the individual components of the composite scores, health measures (hospital admissions and deaths), and indicators of appropriate management of comorbid conditions such as cardiovascular risk factors. Eligible patients will be identified and outcomes measured using electronic medical records.

DETAILED DESCRIPTION:
Long-lasting lung diseases like asthma and chronic obstructive lung disease (COPD) - collectively called chronic respiratory disease (CRD) - place a heavy and growing burden on people living in low and middle income countries. Many of them could be healthier if their disease was accurately diagnosed and correctly treated, but many are not. Doctors and nurses working in primary health care clinic are best placed people to diagnose and treat CRD, especially where local clinics are near and free. But this raises three questions: 1. How to ensure that CRDs get the priority they need in overloaded clinics? 2. How to train clinicians to diagnose and manage CRDs without special test equipment? 3. How to ensure rational evidence-based diagnosis and prescribing for CRD?

The investigators have developed a way of improving primary health care for people who have CRD, who often also have other long term health conditions. It is a patient management tool (PMT), that is, a printed manual of flowcharts taking doctors and nurses from symptoms to diagnoses to treatments, tests or referrals, with advice on how to make decisions along the way about diagnoses, tests, treatments and referrals. They are prompted to think of other diseases and health problems that might be undetected or neglected. The package also includes a method of training known as outreach education. First trainers are trained, then trainers train groups of doctors and nurses at their workplaces, showing them how to use the guidelines, and using their own patients and clinical problems as examples. This outreach training is repeated several times in short sessions. The investigators' research in Africa has shown that this approach can be effective, cost effective, feasible and sustainable. It has been rolled out throughout South Africa and other African countries. But it has have not yet been shown to be effective for this combination of diseases (CRDs together with cardiovascular disease, diabetes, tuberculosis and back pain). The investigators have also not tried or evaluate it in Latin American countries, which have different health systems, and have many more doctors providing primary health care. Now co-investigators in the Brazilian city of Florianopolis have decided to put this educational package in place throughout the city, and have agreed to do so as a randomised controlled trial. This will clearly show whether PACK Brazil is effective, cost effective and feasible under Brazilian conditions.

The core of the research will be the randomised controlled trial. 48 primary care clinics in the city will be randomly chosen either 1) to get the whole package of patient management tool plus training, or 2) only to get the patient management tool (which we expect will make little difference without training). The investigators will compare patients in these two groups of clinics to see the effects of the training. They will use the clinics' electronic medical records to identify about 2000 adults diagnosed with asthma or COPD. After the training starts they will follow these patients up for a year, and assess whether they are being appropriately treated and tested. They will also compare the rates of new diagnoses of asthma and COPD in each clinic, and various health indicators.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic lower respiratory diseases (ICD10: J40-J47) recorded in electronic medical records since January 1st 2010

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1950 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Asthma composite score | During first year of follow-up
  For participants with asthma the composite score will comprise points awarded for: i) a first prescription of an inhaled corticosteroid (ICS) or ICS+ long-acting bronchodilator (LABA) combination, or a change in prescription, stepping up from short acting bronchodilator (SABA) to ICS or from ICS to long acting bronchodilator(LABA)+ICS combination; or stepping down from LABA+ICS to ICS, or from ICS to SABA (scoring one point if at least one of these occurs); and ii) request for spirometry (one point). The composite score will be the sum of these points, and will thus range from 0-2. The composite scores for each patient for all visits during the year will be averaged.
COPD composite score | During first year of follow-up
  For participants with COPD the composite score with comprise points awarded for: i) a first prescription of SABA, ICS, or ICS+LABA; or a change in prescription, stepping up from SABA to LABA or LABA to ICS+LABA, or stepping down from LABA+ICS to LABA, or from LABA to SABA (scoring one point if at least one of these occurs) and ii) request for spirometry (one point). The composite score will be the sum of these, and will thus also range from 0-2.
Asthma-or-COPD diagnosis rate | During first year of follow-up
  Among all participants aged 18 years and over attending each clinic, the number of patients in whom either asthma or COPD is diagnosed for the first time

SECONDARY OUTCOMES:
Hospital admission rate for asthma | During first year of follow-up
  Hospital admission rate for asthma in each clinic
Hospital admission rate for COPD | During first year of follow-up
  Hospital admission rate for COPD in each clinic
Cardiovascular disease diagnoses | During first year of follow-up
  Number of patients with asthma or COPD in whom cardiovascular disease (ICD10 code I00-I99) is diagnosed for the first time
Diabetes mellitus diagnosis | During first year of follow-up
  Number of patients with asthma or COPD in whom diabetes mellitus (ICD10 code E10-E14) is diagnosed for the first time
Smoking cessation prescriptions | During first year of follow-up
  Number of participants in whom nicotine replacement therapy, nortryptiline, or bupropion are prescribed
CVD risk assessment | During first year of follow-up
  Number of participants in whom blood pressure is recorded, or for whom cholesterol, glucose, or electrocardiogram tests are recorded
Depression diagnosis | During first year of follow-up
  Number of participants in whom depression (ICD10 code F32-F34) is diagnosed for the first time
Depression treatment | During first year of follow-up
  Number of participants in whom medication for depression (tricyclic and related antidepressants, selective serotonin re-uptake inhibitors, and monoamine oxidase inhibitors) is prescribed for the first time
Death | During first year of follow-up
  Number of participants who died

CONTACTS AND LOCATIONS:
Overall Officials: Max Bachmann, MBChB PhD, Principal Investigator — University of East Anglia; Eric Bateman, MBChB MD, Principal Investigator — University of Cape Town; Rafael Stelmach, MD PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Florianopolis City Health Department, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shekar S, Bachmann MO, Bateman ED, Stelmach R, Cruz AA, Zonta R, Pacheco de Andrade M, Zepeda J, Cornick RV, Wattrus C, Georgeu-Pepper D, Anderson LF, Lombard C, Fairall LR. Effects of PACK training on the management of asthma and chronic obstructive pulmonary disease by primary care clinicians during 2 years of implementation in Florianopolis, Brazil: extended follow-up after a pragmatic cluster randomised controlled trial with a stepped-wedge design. BMJ Glob Health. 2024 Oct 28;9(Suppl 3):e013819. doi: 10.1136/bmjgh-2023-013819. PMID 39467591
- [Derived] Bachmann MO, Bateman ED, Stelmach R, Cruz AA, Pacheco de Andrade M, Zonta R, Zepeda J, Natal S, Cornick RV, Wattrus C, Anderson L, Georgeu-Pepper D, Lombard C, Fairall LR. Effects of PACK guide training on the management of asthma and chronic obstructive pulmonary disease by primary care clinicians: a pragmatic cluster randomised controlled trial in Florianopolis, Brazil. BMJ Glob Health. 2019 Dec 16;4(6):e001921. doi: 10.1136/bmjgh-2019-001921. eCollection 2019. PMID 31908865
- [Derived] Bachmann MO, Bateman ED, Stelmach R, Cruz AA, Pacheco de Andrade M, Zonta R, Zepeda J, Natal S, Cornick R, Wattrus C, Anderson L, Lombard C, Fairall LR. Integrating primary care of chronic respiratory disease, cardiovascular disease and diabetes in Brazil: Practical Approach to Care Kit (PACK Brazil): study protocol for randomised controlled trials. J Thorac Dis. 2018 Jul;10(7):4667-4677. doi: 10.21037/jtd.2018.07.34. PMID 30174920